CLINICAL TRIAL: NCT05870423
Title: Improving Peptide Receptor Radionuclide Therapy With PARP Inhibitors
Acronym: PRRT-PARPi
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Morticia N. Becx, coordinating investigator, Erasmus Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL79259.078.21
Record Dates: First submitted 2023-04-06; First posted 2023-05-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors; Peptide Receptor Radionuclide Therapy
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: 3+3 dose-escalation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PRRT + olaparib 100mg q.d. (Experimental): administration of the standard therapy of 7.4GBq 177lu-dotatate with the additional study medication olaparib 100mg q.d.
  Interventions: Drug: olaparib
- PRRT + olaparib 100mg b.i.d. (Experimental): administration of the standard therapy of 7.4GBq 177lu-dotatate with the additional study medication olaparib 100mg b.i.d.
  Interventions: Drug: olaparib
- PRRT + olaparib 200mg b.i.d. (Experimental): administration of the standard therapy of 7.4GBq 177lu-dotatate with the additional study medication olaparib 200mg b.i.d.
  Interventions: Drug: olaparib
- PRRT + olaparib 300mg b.i.d. (Experimental): administration of the standard therapy of 7.4GBq 177lu-dotatate with the additional study medication olaparib 300mg b.i.d.
  Interventions: Drug: olaparib

INTERVENTIONS:
Drug: olaparib — 18 days olaparib during each cycle of PRRT
  Other Names: Lynparza

SUMMARY:
This is a phase 1 dose-escalation study to determine the maximum tolerated dose of the PARP inhibitor olaparib in combination with PRRT in patients with a well-differentiated advanced gastroenteropancreatic NET (GEP NET), progressive after PRRT. As secondary objectives, efficacy, pharmacokinetics and biomarker response will be investigated.

DETAILED DESCRIPTION:
Rationale:

Peptide receptor radionuclide therapy (PRRT) with the beta-emitting radiopharmaceutical 177Lutetium-DOTA-Tyr3,octreotate (177Lu-DOTATATE) is an effective and safe treatment option for patients with metastatic neuroendocrine tumors (NETs). In advanced NET patients, 177Lu-DOTATATE has been proven to secure long-term survival in several large retrospective series and was superior to high-dose somatostatin analogs in a randomized phase 3 clinical trial, with a 79% decrease in the risk of progression or death. However, objective response rates are limited and fewer than 1% of the patients can achieve complete response following PRRT. Administering a higher cumulative dose than currently applied will induce more toxicity in healthy tissues and probably will be detrimental to patients. Therefore, adaptations to the currently applied PRRT regimen are needed.

The repair of PRRT-induced DNA damage constitutes a viable target to enhance its antitumor effects. In a number of preclinical models, inhibitors of the enzyme poly ADP ribose polymerase (PARP), essential for repair of single-strand DNA breaks, have been shown to improve the cytotoxic effects of PRRT without signs of added toxicity. Various PARP inhibitors are registered for the treatment of human cancers, such as ovarian cancer, and BRCA- or homologous repair deficiency (HRD)-dependent prostate and pancreatic cancer and are under investigation in several clinical trials as radiosensitizer. Based on preclinical in vitro and in vivo data, we hypothesize that PARP inhibitors can potentiate radiation-induced tumor cell death in patients treated with PRRT. This therapeutic combination has not been studied in human subjects before.

Objective:

To determine the maximum tolerated dose (MTD) of the PARP inhibitor olaparib in combination with PRRT in patients with a well-differentiated advanced NET, progressive after PRRT.

Study design:

Phase I dose escalation, single arm, prospective single center study.

Study population:

Patients with locally advanced or metastatic NETs that have progressive disease according to RECIST v1.1 following initial or salvage PRRT and are considered for two additional PRRT cycles of standard 7.4 GBq each.

Intervention:

Patients eligible for retreatment with PRRT will receive the PARP inhibitor olaparib starting 3 days before each dose of 7.4 GBq 177Lu-DOTATATE until 2 weeks thereafter. The dose of olaparib will be increased from 100 mg q.d. to 300 mg b.i.d. in subsequent patients in 4 preplanned dose escalation steps. In case of unexpected toxicity at the start dose, a de-escalation step to 50 mg q.d. is allowed. The study is performed according to the classic phase I 3+3 dose escalation design with initially 3 patients per dose level. If no dose-limiting toxicity (DLT) is observed in 3 consecutive patients, the dose will be increased to the next planned dose-level. In case of 1 DLT, inclusion of up to 3 additional patients at the same dose is pursued, after which dose escalation can follow if no additional DLT is observed. In case of ≥2/6 DLTs at a given dose level, further dose escalation will be stopped and an additional 3 patients will be treated at the next lower dose level in order to establish a recommended phase II dose (R2PD) for further testing.

Main study parameters/endpoints:

Primary endpoints:

* Incidence and severity of adverse events according to CTCAE v5.0
* Determination of the MTD of olaparib in combination with standard dose PRRT

Secondary endpoints:

* Progression-free and overall survival
* Response rate
* Olaparib pharmacokinetic parameters
* Pharmacokinetic/-dynamic influence of olaparib on 177Lu-DOTATATE
* Measurement of antitumor effects in freshly acquired tumor biopsies

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced or metastatic, well-differentiated (grade 1, 2 or 3) NET.
* Disease progression based on RECIST v1.1 following initial or salvage treatment with PRRT with 177Lu-DOTATATE with a progression free interval of at least 12 months since first cycle of previous administration of PRRT or with no suitable systemic alternative treatment options.
* The patient is eligible for two cycles of salvage PRRT.
* Measurable disease according to RECIST v1.1 on CT/MRI.
* Confirmed presence of somatostatin receptors on all target lesions on CT/MRI, based on positive uptake on a 68Ga-DOTATATE/-TOC/-NOC PET-CT/MRI scan.
* Age ≥ 18 years.
* Karnofsky Performance Score (KPS) > 60.

Exclusion Criteria:

* Hb concentration <6.2 mmol/L; white blood cell count <3x109/L; platelets <100x109/L; neutrophil count <1.5x109/L.
* Renal insufficiency defined as a creatinine clearance <50 mL/min, measured in 24-hour urine collection.
* Liver function or enzyme abnormalities defined as a total bilirubin >3 x ULN, Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 x ULN or serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
* Pregnancy, lactation and inability to comply with effective means of contraception in females of child-bearing age.
* Neuroendocrine carcinoma of any origin.
* Any surgery, radioembolization, chemoembolization, chemotherapy and radiofrequency ablation within 12 weeks prior to inclusion in the study. Interferons, everolimus, sunitinib or other systemic therapies within 4 weeks prior to inclusion in the study.
* Uncontrolled congestive heart failure (NYHA II, III, IV).
* Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with the completion of the study.
* Prior external beam radiation therapy to more than 25% of the bone marrow.
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and proven no evidence of recurrence for 5 years.
* Patients who use a strong CYP3A4 inhibitor within 1 week before start of the treatment or a CYP3A4 inducer within 4 weeks before start of the treatment.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Known allergy or intolerance for the (non-)investigational drugs.
* Inability to provide informed consent.
* End of life care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 3 years
  Incidence and severity of adverse events according to CTCAE v5.0
Maximum tolerated dase | 3 years
  Determination of the MTD of olaparib in combination with standard dose PRRT

SECONDARY OUTCOMES:
Survival rates | 3 years
  Progression-free and overall survival
Best response | 3 years
  Response rate
Antitumor effects | 3 years
  Measurement of antitumor effects in freshly acquired tumor biopsies. DNA damage, transcriptomics and PARylation will be measured in blood and tumor biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided